CLINICAL TRIAL: NCT05289856
Title: A Phase II, Open-label, Multicenter Trial to Investigate the Clinical Activity and Safety of Cabozantinib in Combination With Avelumab in Patients Refractory to Standard Chemotherapy With Advanced Neuroendocrine Neoplasias G3 (NEN G3).
Brief Title: Cabozantinib in Combination With Avelumab in Patients Refractory to Standard Chemotherapy With Advanced Neuroendocrine Neoplasias G3 (NEN G3)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Ipsen (Industry); Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Matthias M. Weber, Professor, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaboAveNEC; 2021-000986-34 (EudraCT Number)
Record Dates: First submitted 2022-03-07; First posted 2022-03-22 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cancer
Keywords: neuroendocrine neoplasias (NEN); NET G3; NEC G3; avelumab; cabozantinib
MeSH Terms: conditions — Neoplasms | interventions — cabozantinib; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination of Avelumab and Cabozantinib (Experimental): 800 mg Avelumab every 2 weeks and 40 mg Cabozantinib daily
  Interventions: Drug: combination of Avelumab and Cabozantinib

INTERVENTIONS:
Drug: combination of Avelumab and Cabozantinib — Cabozantinib 40 mg daily PO in combination with Avelumab at a dose of 800 mg as a 1h intravenous (i.v.) infusion every two weeks (q2w) until disease progression (PD), unacceptable toxicity, or any criterion for treatment withdrawalis met, for a maximum of 12 months
  Other Names: Bavencio; Cabometyx

SUMMARY:
The purpose of the CaboAveNEC trial is to investigate the clinical activity and safety of Cabozantinib in combination with avelumab in patients refractory to standard chemotherapy with advanced neuroendocrine neoplasias G3 (NEN G3).

DETAILED DESCRIPTION:
According to the WHO classification of 2010, Neuroendocrine neoplasms (NEN) are graded according to the Ki67 proliferation index and grouped into neuroendocrine Tumors (NET) Grade 1 (NET G1, Ki67 <3%), NET G2 (Ki67 3-20%), and neuroendocrine Carcinomas (NEC) (G3, Ki67 >20%). However, since the WHO 2017/2019 classification the group of gastrointestinal neuroendocrine tumors with a Ki67 ≥20% (NEN G3) is subdivided according to their morphology into highly proliferative differentiated NET G3 and poorly differentiated high grade neuroendocrine Carcinomas (NEC G3, Ki67 > 20%), which - depending on their morphology - are subdivided into small cell as well as large cell NECs. The vast majority (60-90%) of patients with high grade NEC are metastasized at the time of diagnosis with distant metastases present in approximately two third of the patients.

The prognosis of patients with metastatic NEN G3 is poor, and median overall survival has been reported to be 5 months with a 2-year survival rate of 11 % in the SEER data base for gastrointestinal NEC. In two large series of GEP-NEC, median survival was 12-19 months for patients with best available therapy (mainly platinum based chemotherapy) and as short as 1 month for those receiving only best supportive therapy. In contrast to the "classical" undifferentiated NEC G3 with a poorly differentiated morphology and a Ki 67 > 55%, NET G3 typically do not respond as well to a platinum based chemotherapy but a have a somewhat better prognosis with a 4-months longer median survival as compared to classical NEC G3. Therefore, according to current guidelines other treatment options like temozolomide based chemotherapy may be considered as a first line therapy in patients with differentiated "NET G3".

There is a strong and unmet medical need for a novel and effective second line treatment option for these highly aggressive and rapidly progressing tumors.

Considering the lack of any other established therapeutic option and the very limited efficacy of alternative second or third line chemotherapy in patients with NEN G3 who are progressive after a first-line chemotherapy, the availability of a novel therapeutic option with a significant clinical benefit (SD; PR; CR) in at least 40 % of the patients and with tolerable side effects would represent an important and clinical highly relevant break through in the treatment of these aggressive tumors.

Avelumab is a fully human antibody that binds PD-L1 and blocks the interaction between PD-L1 and PD-1. This removes the suppressive effect of PD-L1 on anti-tumor CD8+ T cells, resulting in restoration of cytotoxic T cell response.

In the ongoing phase II trial of the investigator (AveNEC, EudraCT No: 2016-004373-40), which is the largest immunotherapy trial in patients with NEN G3, the clinical activity and safety of the PD-L1 inhibitor avelumab is evaluated in 60 patients with advanced, metastatic NEN G3 progressive after chemotherapy. According to the interim analysis presented at ASCO 2019 a clinically meaningful response was seen in 27 % of patients with a significant longer progression free survival (mean PFS 33.5 vs 7.7 weeks) and overall survival (> 60 weeks mean not reached vs 22.4 weeks) as compared to the non-responders.

Cabozantinib is a multikinase inhibitor of MET, VEGFR, AXL and RET which is currently being used very successfully in medullary thyroid carcinoma (MTC), which is a differentiated neuroendocrine neoplasia, in advanced renal cell carcinoma (RCC) and hepatocellular carcinoma (HCC).

In addition to its TKI activity, there is strong evidence that Cabozantinib modulates the tumor immune microenvironment leading to a synergistic efficacy in combination with a checkpoint inhibitor therapy.

There is an especially strong rationale for a combination therapy of the potent antiangiogenic TKI Cabozantinib with the checkpoint inhibitor Avelumab in NEN G3. Both drugs have demonstrated efficacy and safety in combination therapy studies of a checkpoint inhibitor and an antiangiogenic TKI in a variety of tumors and both drugs in monotherapy have shown clinical relevant antitumor efficacy in NEN.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically proven neuroendocrine neoplasia NEN G3 (WHO 2010/2019)
3. One block or 20 slides (cut at 4 microns) of archival tumor tissue to perform central pathological review and biomarker assessment and for translational research
4. No curative option available
5. Progression within 9 months before study initiation and after at least one chemotherapy (platinum based chemotherapy or STZ/TEM/DTIC based chemotherapy)
6. Presence of measurable disease as per RECIST1.1 criteria
7. Adequate organ and bone barrow functionn:

   1. Hematologic: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused)
   2. Hepatic: total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 × ULN for subjects with documented metastatic disease to the liver)
   3. Renal: estimated creatinine clearance ≥ 60 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)
8. Pregnancy and contraception:

   1. Pregnancy test: Negative serum or urine pregnancy test at screening for women of childbearing potential.
   2. Contraception: Women of child-bearing potential (WOCBP) and men who are able to father a child, willing to be abstinent or use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at informed consent, for the duration of study participation and for at least 30 days for female and 90 days for male patients after last dose of avelumab and at least for 4 months after last dose of cabozantinib
9. ECOG Performance Status 0 - 1
10. Life expectancy of at least 12 weeks according to the assessment of the investigator
11. Written informed consent: Signed and dated informed consent of the subject must be available before start of any specific trial procedures
12. Ability of subject to understand nature, importance and individual consequences of clinical trial.

Exclusion Criteria:

1. Merkel Cell carcinoma (MCC) or small cell lung cancer (SCLC)
2. Typical or Atypical Carcinoid of the lung with a Ki67 < 20%
3. Prior therapy with any TKI or immune therapy
4. Neuroendocrine neoplasias that are potentially curable by surgery
5. Major surgery within 4 weeks before first dose of study medication. Complete wound healing must be observed at least 10 days prior to enrollment.
6. Patients who are at increased risk for severe haemorrhage
7. TACE, TAE, SIRT or PRRT within 8 weeks before first dose of study medication
8. Patients pretreated with Interferon as last treatment line prior to study entry
9. Concurrent anticancer treatment after start of trial treatment (e.g., cyto¬reductive therapy, TKI therapy, mTOR inhibitor therapy, radiotherapy [with the exception of palliative radiotherapy], immune therapy, or cytokine therapy except for erythropoietin or use of any investigational drug).
10. Concurrent treatment with strong inducers of cytochrome P450 3A4 (eg, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's wort) and strong inhibitors of cytochrome P450 3A4 (eg, ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, and ritonavir), warfarin (due to its high protein bound)
11. Immunosuppressants: Current use of immunosuppressive medication, EXCEPT for the following:

    1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
    2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
12. Prior organ transplantation, including allogeneic stem cell transplantation
13. Active infection requiring systemic therapy
14. HIV/AIDS: Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
15. Hepatitis: Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
16. Active SARS-CoV-2 infection (detected via positive PCR test)
17. Autoimmune disease: Severe active autoimmune disease that requires immunomodulatory therapy. Patients with diabetes type I, vitiligo, psoriasis, autoimmune thyroid disease not requiring immunosuppressive treatment are eligible.
18. Persisting toxicity related to prior therapy (NCI CTCAE v.5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
19. Pregnancy or lactation
20. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
21. Vaccination: Vaccination within 4 weeks before the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines.
22. Hypersensitivity to study drugs: Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3) and lactose contained in cabozantinib tablets
23. Cardiovascular disease: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), uncontrolled arterial hypertension or serious cardiac arrhythmia requiring medication.
24. Clinical significant hematemesis or hemoptysis
25. Medical or psychological conditions that would jeopardise an adequate and orderly completion of the trial
26. Patients, who are legally institutionalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR: CR, PR, SD) | 16 weeks
  Disease control rate (DCR: CR, PR, SD) according to iRECIST after 16 weeks from start of treatment until documented disease progression (PD)

SECONDARY OUTCOMES:
Disease control rate (DCR: CR, PR, SD) | week 8, week 24, week 48
  Disease control rate (DCR: CR, PR, SD) according to iRECIST
Objective response rate (ORR) | week 8, week 16, week 24, week 48
  Objective response rate (ORR) according to iRECIST
Best overall response (BOR) | week 8, week 16, week 24, week 48
  Best overall response (BOR) according to iRECIST
Duration of disease control (DDC) | week 48
  Duration of disease control (DDC) according to iRECIST
Time to response (TTR) | week 48
  Time to response (TTR) according to iRECIST
Progression-free survival time (PFS) | week 48
  Progression-free survival time (PFS) according to iRECIST
Evaluation of tumor response according to RECIST1.1 | week 8, week 16, week 24, week 48
  Evaluation of tumor response according to RECIST1.1
Overall survival (OS) | week 48, week 96
  Overall survival (OS)
Quality of life (QoL) | week 8, week 16, week 24, week 48
  Quality of life (QoL) assessed by European Organisation for Research and Treatment of Cancer Quality of life questionnaire (EORTC QLQ-C30); Scale 0 - 100; higher levels indicate better quality of life
Adverse events | week 48
  Number, severity, and duration of treatment-emergent AEs according to NCI-CTCAE v5.0
Dose change of study drugs | week 48
  Dose change of study drugs
Treatment interruption or termination | week 48
  Treatment interruption or termination of study drugs due to adverse events

OTHER OUTCOMES:
Correlation of the primary and secondary endpoints with the differentiation of the NEN G3 | week 8, week 16, week 24, week 48
  Correlation of the primary and secondary endpoints with the differentiation of the NEN G3 (NET G3 vs NEC) and tumor immune microenvironment (e.g. PD-L1 expression, TIL)
Comparison of the efficacy and tolerability of the combination treatment with Cabozantinib and Avelumab to the monotherapy with Avelumab | week 8, week 16, week 24, week 48
  Comparison of the efficacy and tolerability of the combination treatment with Cabozantinib and Avelumab to the monotherapy with Avelumab in the AveNEC trial (EudraCT No.: 2016-004373-40)
Evaluation of tumor growth rate (TGR) | week 8, week 16, week 24, week 48
  Evaluation of tumor growth rate (TGR): TGR is the percentage change in tumour volume over one month

CONTACTS AND LOCATIONS:
Overall Officials: Matthias M Weber, MD, Principal Investigator — Universitätsmedizin der Johannes Gutenberg-Universität Mainz, I. Medizinische Klinik und Poliklinik, Abteilung Endokrinologie und Stoffwechselkrankheiten, D-55131 Mainz, Germany
Locations (2):
- Germany (2):
  - Nationales Centrum für Tumorerkrankungen, Universitätsklinikum Heidelberg, Heidelberg
  - I. Medizinische Klinik und Poliklinik, Endokrinologie und Stoffwechselerkrankungen, Universitätsmedizin Mainz, Mainz

IPD SHARING:
Plan to Share IPD: No